CLINICAL TRIAL: NCT02571231
Title: Pilot Study: High Flow Ventilation With Volume Guarantee
Brief Title: High Flow Ventilation With Volume Guarantee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OsloUH_bogland
Record Dates: First submitted 2015-09-28; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Rds; Pulmonary Hypertension; Meconium Aspiration Syndrome
MeSH Terms: conditions — Acute Lung Injury; Hypertension, Pulmonary; Meconium Aspiration Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HFV+vg (Experimental): volume guarantee given
  Interventions: Device: HFV + and - VG
- HFV-VG (Experimental): Volume guarantee not given
  Interventions: Device: HFV + and - VG

INTERVENTIONS:
Device: HFV + and - VG — High frequency ventilation with and without volume guarantuee

SUMMARY:
The trial is a pilot study performed in the NICU's at Oslo University Hospital and Haukeland University Hospital preparing a multi-center randomized, controlled unblinded cross-over study, comparing high frequency ventilation (HFV) with and without volume guarantee (VG).

DETAILED DESCRIPTION:
HFV is a way to deliver mechanical breathing support to patients with respiratory failure applied in Neonatal Intensive Care Units (NICU's). In some NICU's, this mode of ventilation is applied when conventional ventilation fails, whereas in other units HFV is used as the primary ventilation mode.

HFV is a ventilator mode where high frequency pressure changes, typically 6-12 per second (6 - 12 Hertz (Hz)), is used to exchange air between the lungs (alveoli) and the ventilator tubing.

Concerns have been raised regarding fluctuating PCO2 values in babies receiving HFV. It is believed that stable normocapnia (normal PCO2 values) as opposed to hyper- and hypocapnia is associated to better short and long-term outcomes.

In conventional ventilator modes, CO2 diffusion is a function of the product from volume per breath (Vt) and the frequency (f) of breathing (Vt*f = minute volume (MV)). In HFV the CO2 diffusion is a function of a product from the small tidal volumes generated (Vthf) squared, and the oscillation frequency (Hz) delivered by the ventilator (vthf2 * F=DCO2). The small tidal volumes are being adjusted by altering the pressure range (amplitude) and the frequency by which pressure changes is generated. One challenge in using HFV has been unwanted fluctuations in PCO2 values, which has been shown to be associated with clinical important complications, in particular cerebral hemorrhages. In order to avoid substantial fluctuation in PCO2 a meticulous adjustment of the amplitude is required.

Modern neonatal ventilators now offer the ability to automatically adjust the amplitude of the high frequency breaths to obtain a stable high frequency tidal volume. The ventilator measures the Vthf and increase or decrease the power of each breath to obtain the set Vthf. This mode is called high frequency ventilation with volume guarantee (HFV+VG).

Automatically adjustment of the amplitude is a novel option in high frequency ventlators and has not been studied in randomized trials.

This study will investigate compare HFV with and without VG. Patients treated with HFV will be randomized to conventional HFV or HFV+VG. After 24 hours the mode will be changed to HFV+VG for those starting on HFV and to HFV for those starting on HFV+VG for 24 hours. After the trial period of 24 x 2 hours - the HFV mode will be at the clinician's preference.

To compare the efficiency of both modes of HFV, measured PCO2 values, oxygen need and variables from the ventilator will be sampled. These variables describe the effort from the ventilator (frequency, amplitude) as well as variables associated with gas exchange in the lungs (Vthf, DCO2).

ELIGIBILITY:
Inclusion Criteria:

* all neonates in need of high frequency ventilator

Exclusion Criteria:

* neonates expected to need high frequency ventilator less than 48 hours because of planned surgery etc

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
stability of High Frequency Tidal volumes | during study, ie. 48 hours.
  HFVVt are measured by ventilator.
Stability of CO2 measurements | during study, ie. 48 hours.
  Measured CO2 values will be measured as usual
frequency of needed manual adjustments on the ventilator | during study, ie 48 hours
  Adjustments made on ventilator will be automatically sampled by the ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn e Ogland, md dr philos, Principal Investigator — Oslo University Hospital